CLINICAL TRIAL: NCT00677222
Title: A Phase I, Multicenter, Dose-Escalation Trial Evaluating the Safety of Allogeneic AMI MultiStem® in Patients With Acute Myocardial Infarction
Brief Title: Safety Study of AMI MultiStem® to Treat Heart Attacks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Healios K.K. (Industry)
Collaborators: PPD Development, LP (Industry); Angiotech Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMI-07-001
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction, Heart Attack
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Treatment arm
  Interventions: Biological: AMI MultiStem®
- 2 (No Intervention): Registry Arm -standard of care

INTERVENTIONS:
Biological: AMI MultiStem® — AMI MultiStem® administered via catheter into peri-vascular space of the target vessel, 2-5 days post PCI. There will be 3 dose escalation cohorts, 6 patients per cohort.
  Arms: 1

SUMMARY:
The purpose of this study is to determine if escalating doses of AMI MultiStem® delivered by catheter can safely be given to patients that have had a recent heart attack treated with stent implantation.

DETAILED DESCRIPTION:
The mortality rates associated with acute myocardial infarction (AMI) have significantly decreased over the past 2 decades. Beginning first with thrombolytic therapy for AMI, and more recently with growing acceptance and availability of primary percutaneous coronary intervention (PCI) for ST-elevation AMI, the mortality rates of this devastating ischemic event have decreased from almost 15% in clinical trials in the late 1980's to <5% in recent primary percutaneous coronary intervention trials. Though AMI-related mortality has been reduced, AMI survival is often accompanied by significant loss of function that may lead to subsequent treatments, congestive heart failure (CHF) and reduction in quality of life. A cell therapy that could reduce the damage associated with AMI and positively affect heart function would provide substantial benefits to the AMI patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex 18-85 years of age
* Women of childbearing potential or less than 2 years postmenopausal agree to use of adequate contraception during the study
* Patients with the first time diagnosis of ST elevation myocardial infarction
* Acute myocardial infarction (ST elevation in at least two leads >0.2 mV in V1, V2 or V3 or >0.1 mV in other leads), treated by one of the following: either
* Acute PCI with stent implantation
* With thrombolysis within 12 hr of symptom onset followed by PCI with stent implantation within 24 hr after Thrombolysis
* Maximal creatine kinase elevation >400 U/l with significant membrane-bound fraction (>6%)or troponin >2X ULN
* Decreasing levels of CK/CK-MB or troponin following reperfusion
* Successful acute PCI/stent implantation (residual stenosis visually <30% and TIMI flow >2). Absence of severe disorder of the microcirculation (e.g. pulsatile flow pattern, systolic flow reversal) at the time of administration of the trial therapy
* Significant regional wall motion abnormality in left ventricular angiogram or transthoracic echocardiogram ≤48 hours post PCI
* LVEF between 30 and 45% by LV gram after the primary PCI or transthoracic echocardiogram ≤48 hours post PCI
* Willing and able to comply with the scheduled visits, treatment, laboratory tests and other study related procedures.
* Signed informed consent

Exclusion Criteria:

* Prior cardiovascular history
* Mechanical complications of the index acute myocardial infarction including but not limited to rupture of the mitral valve with resultant development of mitral regurgitation, rupture of the left ventricular free wall and rupture of the interventricular septum
* Pregnant or lactating
* Known allergy to contrast agents
* Known allergy or religious objections to bovine or porcine products
* History of malignancy of any type except non-melanoma skin cancer
* Presence of major hematological conditions or laboratory abnormalities (low hemoglobin (<10 gm/dl), - WBC (<3,000 cells/mm2) or platelet count (<100,000 cells/mm3))
* Prothrombin time (PT) > 1x ULN
* Partial thromboplastin time (PTT) > 1x ULN
* Presence of chronic systemic inflammatory disorders that requires ongoing therapy
* Previous autologous, allogeneic bone marrow or peripheral stem cell transplant
* Prior solid organ transplantation
* Immune system compromise including but not limited to history of human immunodeficiency virus (HIV), hepatitis B (HBV) and hepatitis C (HCV) infection.
* Prior participation in any other study involving investigational pharmacological agents(s), devices or marketed products within 30 days prior to planned AMI MultiStem® administration
* Life expectancy of six months or less
* Current alcohol or substance abuse
* Ongoing systemic infection
* Renal function: Serum creatinine >2 mg/dL or creatinine clearance ≤50 mL/min
* Hepatic function: Screening ALT and AST ≥3x upper limit of normal for the laboratory or total bilirubin ≥2.0 mg/dL (exception: acceptable if patient is identified with pre existing condition e.g. Gilbert's disease that will contribute to baseline elevations of bilirubin)
* Other serious medical or psychiatric illness that, in the investigator's opinion, would not permit the patient to be managed according to the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events during the first 24 hours after administration of AMI MultiStem® and post acute adverse events up to 30 days following AMI | 30 days

SECONDARY OUTCOMES:
Evaluation of longer term safety and cardiac function over 12 months following AMI | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Penn, MD, Principal Investigator — The Cleveland Clinic; Warren Sherman, MD, Principal Investigator — Columbia University
Locations (7):
- United States (7):
  - Cardiology PC, Birmingham, Alabama
  - The Care Group, Indianapolis, Indiana
  - Henry Ford Hospital, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Metro Health, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Hamot Medical Center, Erie, Pennsylvania

REFERENCES:
- [Derived] Penn MS, Ellis S, Gandhi S, Greenbaum A, Hodes Z, Mendelsohn FO, Strasser D, Ting AE, Sherman W. Adventitial delivery of an allogeneic bone marrow-derived adherent stem cell in acute myocardial infarction: phase I clinical study. Circ Res. 2012 Jan 20;110(2):304-11. doi: 10.1161/CIRCRESAHA.111.253427. Epub 2011 Nov 3. PMID 22052917